CLINICAL TRIAL: NCT06925737
Title: A Phase 3, Open-label Study of Ifinatamab Deruxtecan Versus Docetaxel in Participants With Metastatic Castration-Resistant Prostate Cancer (mCRPC) (IDeate-Prostate01)
Brief Title: A Clinical Study of Ifinatamab Deruxtecan (I-DXd) in People With Metastatic Prostate Cancer (MK-2400-001)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2400-001; U1111-1312-2498 (Registry Identifier: UTN); 2024-517423-40-00 (Registry Identifier: EU CT)
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer; Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Prednisone; Prednisolone; prednisolone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- I-DXd (Experimental): Participants receive I-DXd 12mg/kg every 3 weeks (q3w)
  Interventions: Drug: Ifinatamab deruxtecan
- Docetaxel (Active Comparator): Participants receive docetaxel 75 mg//m^2 q3w and prednisone 10 mg/day or per approved product label
  Interventions: Drug: Docetaxel; Drug: Prednisone

INTERVENTIONS:
Drug: Ifinatamab deruxtecan — Administered via intravenous (IV) infusion every 3 weeks (q3W) until disease progression, unacceptable adverse events (AEs), or other cessation of treatment
  Other Names: I-DXd; MK-2400
  Arms: I-DXd
Drug: Docetaxel — Administered via IV infusion q3W until disease progression, unacceptable adverse events (AEs), or other cessation of treatment
  Arms: Docetaxel
Drug: Prednisone — Oral tablet administered once per day or per approved product label
  Other Names: Prednisone acetate; Prednisolone; Prednisolone acetate
  Arms: Docetaxel

SUMMARY:
Researchers are looking for new ways to treat metastatic castration-resistant prostate cancer (mCRPC). Researchers have designed a study medicine called ifinatamab deruxtecan (also called I-DXd or MK-2400) to treat mCRPC. The goal of this study is to learn if people who receive I-DXd live longer overall and live longer without the cancer growing or spreading than people who receive chemotherapy,

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has diagnosis of metastatic castration-resistant prostate cancer (mCRPC)
* Has prostate cancer progression while on androgen deprivation therapy (ADT) (or post bilateral orchiectomy) within 6 months prior to entering the study
* Has received prior treatment with 1 or 2 androgen receptor pathway inhibitor (ARPI) and progressed during or after at least 8 weeks of treatment

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* History of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids
* Has uncontrolled or significant cardiovascular disease
* Has received prior treatment with a taxane-based chemotherapy agent for mCRPC

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1440 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2028-06-26 (Estimated); Study Completion 2031-01-06 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to approximately 36 months
  OS is defined as the time from randomization to death due to any cause.
Radiographic Progression Free Survival (rPFS) | Up to approximately 36 months
  rPFS is defined as the time from randomization to the first documented disease progression per prostate cancer working group (PCWG)-modifed Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 by blinded independent central review (BICR) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Time to First Subsequent Therapy (TFST) | Up to approximately 36 months
  TFST is defined as the time from randomization to initiation of the first subsequent anticancer therapy or death, whichever occurs first.
Objective Response (OR) | Up to approximately 36 months
  The OR is defined as a confirmed complete response (CR) or partial response (PR) per PCWG-modified RECIST 1.1 as assessed by BICR.
Duration of Response (DOR) | Up to approximately 36 months
  For participants who demonstrate confirmed CR or PR, DOR is defined as the time from the first documented evidence of CR or PR until disease progression per PCWG-modified RECIST 1.1 as assessed by BICR or death due to any cause, whichever occurs first.
Time to Pain Progression (TTPP) | Up to approximately 36 months
  TTPP is defined as the time from randomization to pain progression based on the brief pain inventory-short form (BPI-SF) Item 3 "worst pain in 24 hours" and opiate analgesic use (AQA score).
Time to Prostate-specific Antigen (PSA) Progression | Up to approximately 36 months
  Time to PSA progression is defined as the time from randomization to PSA progression. The PSA progression date is defined as the first date that 1) ≥25% increase and ≥2 ng/mL above the nadir which is confirmed by a second value≥3 weeks later if there is PSA decline from baseline, 2) ≥25% increase and ≥2 ng/mL increase from baseline beyond 12 weeks if there is no PSA decline from baseline.
PSA Response | Up to approximately 36 months
  PSA response rate is defined as the proportion of participants in the analysis population who have a PSA reduction of ≥50% from baseline with a consecutive confirmation assessment at least 3 weeks later per PCWG criteria
Time to First Symptomatic Skeletal-related Event (SSRE) | Up to approximately 36 months
  Time to first SSRE is defined as the time from randomization to the first occurrence of any of the following symptomatic skeletal-related events:
  1. use of EBRT to prevent or relieve skeletal symptoms,
  2. new symptomatic pathologic bone fracture (vertebral or non-vertebral),
  3. spinal cord compression,
  4. a tumor-related orthopedic surgical intervention.
Number of Participants Who Experienced at least One Adverse Event (AE) | Up to approximately 36 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
  An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Number of Participants Who Discontinue Study Treatment Due to an Adverse Event (AE) | Up to approximately 36 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
  An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (263):
- United States (42):
  - Mayo Clinic in Arizona - Phoenix ( Site 0044), Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center ( Site 0049), Duarte, California
  - City of Hope Lennar Foundation Cancer Center ( Site 0059), Irvine, California
  - Moores Cancer Center ( Site 0010), La Jolla, California
  - Cedars-Sinai Medical Center ( Site 0068), Los Angeles, California
  - UCLA Hematology/Oncology - Santa Monica ( Site 0002), Los Angeles, California
  - University of California, Irvine (UCI) Health - UC Irvine Medical Center ( Site 0006), Orange, California
  - Rocky Mountain Regional Veterans Affairs Medical Center ( Site 0053), Aurora, Colorado
  - Yale-New Haven Hospital-Yale Cancer Center ( Site 0050), New Haven, Connecticut
  - The GW Medical Faculty Associates ( Site 0057), Washington D.C., District of Columbia
  - Washington DC Veterans Affairs Medical Center ( Site 0056), Washington D.C., District of Columbia
  - Mayo Clinic in Florida-Mayo Clinic Comprehensive Cancer Center ( Site 0077), Jacksonville, Florida
  - Emory University School of Medicine- Grady Campus ( Site 0103), Atlanta, Georgia
  - Winship Cancer Institute, Emory University ( Site 0003), Atlanta, Georgia
  - University of Illinois at Chicago-University of Illinois Cancer Center ( Site 0063), Chicago, Illinois
  - University of Kentucky Chandler Medical Center ( Site 0048), Lexington, Kentucky
  - Greenebaum Comprehensive Cancer Center ( Site 0021), Baltimore, Maryland
  - Beth Israel Deaconess Medical Center ( Site 0043), Boston, Massachusetts
  - Dana Farber Cancer Institute ( Site 0012), Boston, Massachusetts
  - University of Michigan ( Site 0005), Ann Arbor, Michigan
  - Henry Ford Hospital ( Site 0035), Detroit, Michigan
  - Cancer and Hematology Centers of Western Michigan ( Site 0015), Grand Rapids, Michigan
  - Mayo Clinic in Rochester, Minnesota-Mayo Clinic Comprehensive Cancer Center ( Site 0078), Rochester, Minnesota
  - HealthPartners Cancer Research Center-HealthPartners Frauenshuh Cancer Center ( Site 0032), Saint Louis Park, Minnesota
  - HealthPartners Cancer Center at Regions Hospital ( Site 0052), Saint Paul, Minnesota
  - St. Vincent Frontier Cancer Center-Research ( Site 0037), Billings, Montana
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists - Grand Island ( Site 0076), Grand Island, Nebraska
  - Oncology Hematology West P.C. dba Nebraska Cancer Specialists ( Site 0026), Omaha, Nebraska
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 0016), Hackensack, New Jersey
  - Icahn School of Medicine at Mount Sinai ( Site 0009), New York, New York
  - Great Lakes Cancer Care ( Site 0047), Williamsville, New York
  - The James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive C ( Site 0061), Columbus, Ohio
  - Perelman Center for Advanced Medicine ( Site 0067), Philadelphia, Pennsylvania
  - Abramson Cancer Center - Penn Medicine ( Site 0079), Philadelphia, Pennsylvania
  - Memphis VA Medical Center ( Site 0072), Memphis, Tennessee
  - SCRI Oncology Partners ( Site 0074), Nashville, Tennessee
  - UT Southwestern Medical Center ( Site 0039), Dallas, Texas
  - University of Texas-MD Anderson Cancer Center ( Site 0055), Houston, Texas
  - Blue Ridge Cancer Care ( Site 0024), Roanoke, Virginia
  - VA Puget Sound Health Care System ( Site 0054), Seattle, Washington
  - Fred Hutchinson Cancer Center ( Site 0060), Seattle, Washington
  - University Hospital and UW Health Clinics ( Site 0065), Madison, Wisconsin
- Argentina (9):
  - Centro de Oncologia e Investigacion Buenos Aires COIBA ( Site 0136), Berazategui, Buenos Aires
  - Instituto de Investigaciones Clinicas Mar del Plata ( Site 0129), Mar del Plata, Buenos Aires
  - Instituto Alexander Fleming ( Site 0125), Mar del Plata, Buenos Aires
  - Sanatorio Parque ( Site 0126), Rosario, Santa Fe Province
  - Centro Medico Dra De Salvo ( Site 0132), CABA
  - Fundación CORI para la Investigación y Prevención del Cáncer ( Site 0131), La Rioja
  - Centro Oncologico de Integracion Regional. COIR ( Site 0130), Mendoza
  - Centro de Diagnostico Investigación y Tratamiento Oncológico (CeDIT) ( Site 0135), Salta
  - Instituto San Marcos ( Site 0137), San Juan
- Australia (5):
  - Blacktown Hospital ( Site 0154), Blacktown, New South Wales
  - Macquarie University-MQ Health Clinical Trials Unit ( Site 0151), Macquarie University, New South Wales
  - Gallipoli Medical Research Ltd ( Site 0153), Greenslopes, Queensland
  - Peter MacCallum Cancer Centre ( Site 0152), Melbourne, Victoria
  - Fiona Stanley Hospital ( Site 0155), Murdock, Western Australia
- Austria (3):
  - Ordensklinikum Linz GmbH Elisabethinen-Urologie ( Site 0170), Linz, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH ( Site 0171), Wels, Upper Austria
  - Uniklinikum Salzburg Universitaetsklinik für Innere Medizin III ( Site 0172), Salzburg
- Brazil (6):
  - Hospital Mario Penna ( Site 0179), Belo Horizonte, Minas Gerais
  - Hospital Universitário Evangélico Mackenzie ( Site 0181), Curitiba, Paraná
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre ( Site 0184), Porto Alegre, Rio Grande do Sul
  - Hospital de Base de São José do Rio Preto ( Site 0176), São José do Rio Preto, São Paulo
  - IPITEC ( Site 0189), São Paulo
  - IBCC - Núcleo de Pesquisa e Ensino ( Site 0183), São Paulo
- Chile (2):
  - FALP ( Site 0201), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0200), Santiago, Region M. de Santiago
- China (34):
  - Peking University First Hospital ( Site 1434), Beijing, Beijing Municipality
  - Shanghai General Hospital ( Site 1449), Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chonqing Medical University ( Site 1406), Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Hospital ( Site 1405), Chongqing, Chongqing Municipality
  - The First Affiliated Hospital Of Fujian Medical University ( Site 1452), Fuzhou, Fujian
  - Guangzhou First People's Hospital ( Site 1410), Guangzhou, Guangdong
  - Sun Yat-Sen University Cancer Center ( Site 1467), Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University ( Site 1402), Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center ( Site 1409), Guangzhou, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-Sen University ( Site 1459), Zhuhai, Guangdong
  - Guangxi Medical University Cancer Hospital ( Site 1414), Nanning, Guangxi
  - Henan Cancer Hospital ( Site 1472), Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology ( Site 1424), Wuhan, Hubei
  - Hunan Cancer Hospital ( Site 1411), Changsha, Hunan
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School ( Site 1425), Nanjing, Jiangsu
  - Jiangsu Province Hospital ( Site 1426), Nanjing, Jiangsu
  - Zhongda Hospital Southeast University ( Site 1427), Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University ( Site 1438), Xuzhou, Jiangsu
  - Jilin Province People's Hospital ( Site 1461), Changchun, Jilin
  - The first affiliated Hospital of Xi an Jiaotong University ( Site 1408), Xi'an, Shaanxi
  - Shandong Cancer Hospital ( Site 1421), Jinan, Shandong
  - Shanghai Tenth People's Hospital ( Site 1441), Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center ( Site 1400), Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University ( Site 1430), Shanghai, Shanghai Municipality
  - Shanghai Tongji Hospital ( Site 1412), Shanghai, Shanghai Municipality
  - Renji Hospital Shanghai Jiao Tong University School of Medicine ( Site 1457), Shanghai, Shanghai Municipality
  - First Affiliated Hospital Of Shanxi Medical University ( Site 1460), Taiyuan, Shanxi
  - West China Hospital of Sichuan University ( Site 1451), Chengdu, Sichuan
  - West China Hospital, Sichuan University ( Site 1468), Chengdu, Sichuan
  - The Affiliated Cancer Hospital of Xinjiang Medical University ( Site 1469), Ürümqi, Xinjiang
  - Zhejiang Cancer Hospital ( Site 1447), Hangzhou, Zhejiang
  - The First Hospital of Jiaxing ( Site 1416), Jiaxing, Zhejiang
  - The First Affiliated Hospital of Ningbo University ( Site 1419), Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University ( Site 1437), Wenzhou, Zhejiang
- Colombia (7):
  - Instituto de Cancerología S.A.S ( Site 0234), Medellín, Antioquia
  - Centro Cancerológico del Caribe (CECAC) ( Site 0227), Barranquilla, Atlántico
  - Instituto Nacional De Cancerologia ( Site 0237), Bogotá, Bogota D.C.
  - Clinica Colsanitas S.A, Sede Clínica Universitaria Colombia ( Site 0229), Bogotá, Bogota D.C.
  - Sociedad de Oncología Y Hematología del Cesar S.A.S. ( Site 0228), Valledupar, Cesar Department
  - FUNDACION CTIC CENTRO DE TRATAMIENTO E INVESTIGACION SOBRE CANCER LUIS CARLOS SARMIENTO ANGULO ( Site 0230), Bogota, Cundinamarca
  - Oncologos Del Occidente ( Site 0231), Pereira, Risaralda Department
- Czechia (4):
  - Fakultni nemocnice u sv. Anny v Brne ( Site 0264), Brno, Brno-mesto
  - Masarykuv onkologicky ustav ( Site 0260), Brno, Brno-mesto
  - Fakultni Nemocnice v Motole ( Site 0261), Prague, Praha 5
  - Fakultni nemocnice Olomouc ( Site 0262), Olomouc
- Denmark (4):
  - Herlev and Gentofte Hospital ( Site 0290), Herlev, Capital Region
  - Aalborg Universitetshospital, Syd ( Site 0293), Aalborg, North Denmark
  - Odense Universitetshospital ( Site 0294), Odense, Region Syddanmark
  - Vejle Sygehus ( Site 0291), Vejle, Region Syddanmark
- France (9):
  - Hôpital Foch ( Site 0309), Suresnes, Ain
  - Hôpital Privé Clairval ( Site 0303), Marseille, Bouches-du-Rhone
  - Centre François Baclesse ( Site 0311), Caen, Calvados
  - CHU Besançon ( Site 0305), Besançon, Doubs
  - Centre Hospitalier Universitaire de Nîmes - Institut de Canc-Medical Oncology ( Site 0313), Nîmes, Gard
  - Clinique Francois Chenieux ( Site 0312), Limoges, Haute-Vienne
  - Institut de Cancérologie de Lorraine Alexis Vautrin ( Site 0307), Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHU de Rouen ( Site 0301), Rouen, Seine-Maritime
  - Hôpital Saint-Louis ( Site 0310), Paris, Île-de-France Region
- Germany (8):
  - Studienpraxis Urologie ( Site 0358), Nürtingen, Baden-Wurttemberg
  - Klinikum Stuttgart - Katharinenhospital ( Site 0355), Stuttgart, Baden-Wurttemberg
  - klinikum rechts der isar der technischen universität münchen ( Site 0350), Munich, Bavaria
  - Klinikum Nuernberg Nord ( Site 0353), Nuremberg, Bavaria
  - Urologicum Duisburg ( Site 0361), Duisburg, North Rhine-Westphalia
  - Universitaetsklinikum Schleswig Holstein ( Site 0360), Lübeck, Schleswig-Holstein
  - Charité Universitaetsmedizin Berlin - Campus Mitte ( Site 0352), Berlin
  - Universitaetsklinik Hamburg-Eppendorf ( Site 0351), Hamburg
- Greece (5):
  - Henry Dunant Hospital ( Site 0385), Athens, Attica
  - Metropolitan General Hospital ( Site 0382), Athens, Attica
  - University General Hospital Attikon ( Site 0381), Chaidari Athens, Attica
  - General Oncology Hospital of Kifisia "Agioi Anargyroi" ( Site 0384), Kifissia, Attica
  - Athens Medical Center ( Site 0383), Marousi, Attica
- Guatemala (3):
  - MEDI-K ( Site 0401), Guatemala City
  - Med Clinic ( Site 0403), Guatemala City
  - Onco Go ( Site 0402), Guatemala City
- Hong Kong (2):
  - Queen Mary Hospital ( Site 0415), Hong Kong
  - Tuen Mun Hospital ( Site 0416), New Territories
- Ireland (3):
  - St Vincent's University Hospital ( Site 0441), Dublin, Dublin
  - Cork University Hospital ( Site 0442), Cork
  - Tallaght University Hospital ( Site 0440), Dublin
- Israel (6):
  - Rambam Health Care Campus ( Site 0462), Haifa
  - Meir Medical Center ( Site 0464), Kfar Saba
  - Rabin Medical Center ( Site 0461), Petah Tikva
  - Sheba Medical Center ( Site 0460), Ramat Gan
  - Sourasky Medical Center ( Site 0463), Tel Aviv
  - Yitzhak Shamir Medical Center. ( Site 0466), Ẕerifin
- Italy (9):
  - Fondazione IRCCS Istituto Nazionale dei Tumori ( Site 0500), Milan, Lombardy
  - Istituto Clinico Humanitas ( Site 0504), Rozzano, Milano
  - Istituto Nazionale Tumori Regina Elena ( Site 0507), Rome, Roma
  - Azienda Ospedaliero Universitaria Senese ( Site 0505), Siena, Tuscany
  - Azienda USL 8 di Arezzo ( Site 0503), Arezzo
  - Humanitas Gavazzeni ( Site 0508), Bergamo
  - Azienda Ospedaliero Universitaria Policlinico Riuniti di Foggia ( Site 0510), Foggia
  - Azienda Ospedaliera Santa Maria Terni ( Site 0509), Terni
  - Centro Ricerche Cliniche di Verona ( Site 0506), Verona
- Japan (31):
  - Nagoya University Hospital ( Site 1508), Nagoya, Aichi-ken
  - Toho University Sakura Medical Center ( Site 1503), Sakura, Chiba
  - Ehime University Hospital ( Site 1514), Tōon, Ehime
  - Hospital of the University of Occupational and Environmental Health, Japan ( Site 1510), Kitakyushu, Fukuoka
  - Kurume University Hospital ( Site 1516), Kurume, Fukuoka
  - Sapporo Medical University Hospital ( Site 1501), Sapporo, Hokkaido
  - Hokkaido University Hospital ( Site 1500), Sapporo, Hokkaido
  - Kobe University Hospital ( Site 1511), Kobe, Hyōgo
  - Kanazawa Medical University Hospital ( Site 1507), Kahoku-gun, Ishikawa-ken
  - Shonan Kamakura General Hospital ( Site 1530), Kamakura, Kanagawa
  - Oita University Hospital ( Site 1521), Yufu, Oita Prefecture
  - University of the Ryukyus Hospital ( Site 1519), Ginowan, Okinawa
  - Bell Land General Hospital ( Site 1509), Sakai, Osaka
  - Dokkyo Medical University Saitama Medical Center ( Site 1502), Koshigaya, Saitama
  - Hamamatsu University Hospital ( Site 1520), Hamamatsu, Shizuoka
  - The Jikei University Hospital ( Site 1504), Minato, Tokyo
  - Tokyo Women's Medical University ( Site 1505), Shinjuku, Tokyo
  - Yamaguchi University Hospital ( Site 1522), Ube, Yamaguchi
  - University of Yamanashi Hospital ( Site 1506), Chūō, Yamanashi
  - Harasanshin Hospital ( Site 1517), Fukuoka
  - Kyushu University Hospital ( Site 1515), Fukuoka
  - Gifu University Hospital ( Site 1527), Gifu
  - Hiroshima University Hospital ( Site 1512), Hiroshima
  - Kagoshima University Hospital ( Site 1518), Kagoshima
  - Kagoshima City Hospital ( Site 1528), Kagoshima
  - National Hospital Organization Kumamoto Medical Center ( Site 1524), Kumamoto
  - University Hospital,Kyoto Prefectural University of Medicine ( Site 1525), Kyoto
  - Nagano Municipal Hospital ( Site 1526), Nagano
  - Nagasaki University Hospital ( Site 1523), Nagasaki
  - Niigata Cancer Center Hospital ( Site 1529), Niigata
  - Tokushima University Hospital ( Site 1513), Tokushima
- Mexico (4):
  - Grupo Ollin Care ( Site 0544), Pachuca, Hidalgo
  - CIO - Centro de Inmuno-Oncología de Occidente ( Site 0541), Guadalajara, Jalisco
  - Higiea Oncologia ( Site 0542), Mexico City, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran ( Site 0545), Mexico City, Mexico City
- Netherlands (13):
  - UMC St. Radboud ( Site 0601), Nijmegen, Gelderland
  - Maastricht UMC+ ( Site 0612), Maastricht, Limburg
  - VieCuri Medisch Centrum, locatie Venlo ( Site 0610), Venlo, Limburg
  - Nederlands Kanker Instituut - Antoni van Leeuwenhoek - NKI-AVL ( Site 0602), Amsterdam, North Holland
  - Tergooiziekenhuizen, locatie Hilversum ( Site 0619), Hilversum, North Holland
  - Spaarne Gasthuis - Hoofddorp ( Site 0608), Hoofddorp, North Holland
  - Ziekenhuisgroep Twente, locatie Almelo ( Site 0615), Hengelo, Overijssel
  - Erasmus Medisch Centrum ( Site 0611), Rotterdam, South Holland
  - Franciscus Gasthuis & Vlietland, Locatie Vlietland ( Site 0600), Schiedam, South Holland
  - Haga Ziekenhuis locatie Leyweg ( Site 0607), The Hague, South Holland
  - Meander Medisch Centrum ( Site 0604), Amersfoort, Utrecht
  - Martini Ziekenhuis ( Site 0621), Groningen
  - St. Antonius Ziekenhuis, locatie Utrecht ( Site 0620), Utrecht
- Norway (4):
  - Akershus Universitetssykehus-Onkologisk avdeling ( Site 0650), Lorenskog, Akershus
  - Sykehuset Innlandet HF Gjøvik ( Site 0652), Gjøvik, Oppland
  - St. Olavs Hospital-Kreftklinikken ( Site 0651), Trondheim, Sor-Trondelag
  - Oslo universitetssykehus, Radiumhospitalet ( Site 0653), Oslo
- Peru (3):
  - Hospital Cayetano Heredia ( Site 0667), Lima
  - IPOR Instituto Peruano de Oncología & Radioterapia ( Site 0666), Lima
  - Instituto Neuro Cardiovascular de las Americas ( Site 0668), Lima
- Poland (6):
  - Clinical Research Center Spółka z ograniczoną odpowiedzialnością MEDIC-R Sp.k ( Site 0688), Poznan, Greater Poland Voivodeship
  - Centrum Onkologii im prof Franciszka Lukaszczyka ( Site 0696), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Pratia MCM Krakow ( Site 0692), Krakow, Lesser Poland Voivodeship
  - Mazowiecki Szpital Wojewódzki w Siedlcach-Siedleckie Centrum Onkologii ( Site 0686), Siedlce, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej Curie ( Site 0685), Warsaw, Masovian Voivodeship
  - Pratia Onkologia Katowice ( Site 0693), Katowice, Silesian Voivodeship
- Singapore (2):
  - National Cancer Centre Singapore ( Site 0760), Singapore, Central Singapore
  - Tan Tock Seng Hospital ( Site 0761), Singapore, Central Singapore
- South Africa (5):
  - Cancercare Rondebosch Oncology ( Site 0771), Cape Town, Gauteng
  - Wits Clinical Research ( Site 0776), Johannesburg, Gauteng
  - Wilgers Oncology Centre ( Site 0775), Pretoria, Gauteng
  - Curo Oncology Centre ( Site 0779), Pretoria, Gauteng
  - LIFE GROENKLOOF ( Site 0777), Pretoria, Gauteng
- South Korea (6):
  - Chonnam National University Hwasun Hospital ( Site 0794), Hwasun Gun, Jeonranamdo
  - The Catholic University of Korea St. Mary s Hospital ( Site 0795), Seocho-gu, Seoul
  - Asan Medical Center ( Site 0791), Songpagu, Seoul
  - Ulsan University Hospital ( Site 0793), Donggu, Ulsan-Kwangyokshi
  - Severance Hospital Yonsei University Health System ( Site 0790), Seoul
  - Samsung Medical Center ( Site 0792), Seoul
- Spain (11):
  - Hospital Universitario Marqués de Valdecilla ( Site 0810), Santander, Cantabria
  - CHUS - Hospital Clinico Universitario ( Site 0815), Santiago de Compostela, La Coruna
  - HOSPITAL UNIVERSITARIO PUERTA DE HIERRO MAJADAHONDA ( Site 0811), Majadahonda Madrid, Madrid
  - Hospital General Universitario Gregorio Marañón ( Site 0812), Madrid, Madrid, Comunidad de
  - Hospital del Mar ( Site 0822), Barcelona
  - Hospital Vall D Hebron ( Site 0814), Barcelona
  - Hospital Universitario Reina Sofia ( Site 0816), Córdoba
  - Hospital Lucus Augusti ( Site 0813), Lugo
  - Hospital Universitario Quiron Madrid ( Site 0823), Madrid
  - Hospital Universitario Virgen de Valme ( Site 0819), Seville
  - Fundación Instituto Valenciano de Oncología ( Site 0821), Valencia
- Sweden (4):
  - Skånes Universitetssjukhus Malmö ( Site 0841), Malmo, Skåne County
  - Södersjukhuset ( Site 0844), Stockholm, Stockholm County
  - Karolinska Universitetssjukhuset Solna ( Site 0843), Stockholm, Stockholm County
  - Akademiska sjukhuset-Blod- och tumörsjukdomar ( Site 0840), Uppsala, Östergötland County
- Switzerland (5):
  - Kantonspital Aarau ( Site 0857), Aarau, Canton of Aargau
  - University Hospital Basel ( Site 0859), Basel, Canton of Basel-City
  - Hopitaux Universitaires de Geneve HUG. ( Site 0856), Geneva, Canton of Geneva
  - HFR Fribourg - Hôpital Cantonal ( Site 0858), Fribourg
  - Stadtspital Triemli ( Site 0855), Zurich
- Taiwan (4):
  - National Taiwan University Hospital ( Site 0870), Taiwan, Taipei
  - Chang Gung Medical Foundation - Kaohsiung ( Site 0872), Kaohsiung City
  - Taichung Veterans General Hospital ( Site 0873), Taichung
  - Taipei Veterans General Hospital ( Site 0875), Taipei
- Thailand (2):
  - Faculty of Medicine Siriraj Hospital ( Site 0885), Bangkoknoi, Bangkok
  - Bangkok Metropolitan Administration Medical College and Vajira Hospital ( Site 0887), Dusit, Bangkok
- Turkey (Türkiye) (2):
  - Adana Medical Park Seyhan Hastanesi ( Site 0906), Adana
  - Hacettepe Universitesi Tip Fakultesi ( Site 0895), Ankara

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com